CLINICAL TRIAL: NCT05222724
Title: Efficacy and Safety of the Combination of Ibuprofen and Paracetamol Versus Ibuprofen in Monotherapy in Acute Low Back Pain (LBP)
Brief Title: Efficacy of the Combination of Ibuprofen and Paracetamol in Acute Non-specific Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: TFS Trial Form Support (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 147(Z)WO20157; 2020-005278-86 (EudraCT Number)
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Low Back Pain
Keywords: low back pain; ibuprofen; Paracetamol; Tachifene®
MeSH Terms: conditions — Low Back Pain | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tachifene (Experimental): paracetamol 500 mg/ibuprofen 150 mg FDC, film-coated tablets. Two tablets 3 times daily for 3 days (i.e., every 8 hours ± 1 hour).
  Interventions: Drug: Tachifene
- Brufen (Active Comparator): ibuprofen 600 mg, film coated tablets. One tablet 3 times daily for 3 days (i.e., every 8 hours ± 1 hour).
  Interventions: Drug: Brufen

INTERVENTIONS:
Drug: Tachifene — paracetamol 500 mg/ibuprofen 150 mg FDC, film-coated tablets. Two tablets 3 times daily for 3 days (i.e., every 8 hours ± 1 hour).
  Other Names: paracetamol 500 mg/ibuprofen 150 mg
  Arms: Tachifene
Drug: Brufen — ibuprofen 600 mg, film coated tablets. One tablet 3 times daily for 3 days (i.e., every 8 hours ± 1 hour).
  Other Names: ibuprofen 600 mg
  Arms: Brufen

SUMMARY:
The aim of the present study is to assess the efficacy and safety of paracetamol/ibuprofen Fixed Dose Combination (FDC) compared to ibuprofen in patients with uncomplicated non-specific acute low back pain after a 3-day treatment period.

DETAILED DESCRIPTION:
This is a Phase IV, multicenter, international, open-label, parallel-group study.

The study will be conducted at sites located in Italy, Poland and Hungary. The sites will be outpatient facilities and hospitals. A total of 176 patients are planned to be included in the study This trial will be conducted in accordance with the study protocol, GCPs, Declaration of Helsinki (including up-to-date versions) and applicable regulatory requirements.

The present clinical trial aims to evaluate the efficacy and safety of the combination of 2 tablets of paracetamol 500 mg/ibuprofen 150 mg administered 3 times daily, in the management of patients with acute non-specific Low Back Pain (LBP) condition.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of any ethnic origin between 18 and 64 years of age (limits included).
* Patients with uncomplicated and localized acute low back pain or acute exacerbation of chronic low back pain (not radiating below the gluteal fold), with moderate/severe pain at baseline. Minimum VAS score ≥ 40 mm at screening visit.
* Women of childbearing potential and women with no menses for a period < 12 months must have a negative pregnancy test at Visit 0 and have to agree not to start a pregnancy from the signature of the informed consent up to the Final Visit/Visit 2, using an appropriate birth control method such as combined oestrogen-progestin containing hormonal contraceptives (e.g., oral, injectable, transdermal), progestin-only hormonal contraceptives (e.g., oral, injectable, implantable), intrauterine device (IUD) or Intrauterine hormone-releasing System (IUS) in combination with male condom, bilateral tubal occlusion, vasectomised partner, sexual abstinence. The following definitions will be considered:

  * Woman of childbearing potential (WOCBP): i.e., fertile, following menarche and until becoming post-menopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.
  * A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* Patients legally capable of giving their consent to participate in the study and available to sign and date the written informed consent.

Exclusion Criteria:

* Known hypersensitivity or allergy to the active ingredients and/or to any component of the study medications.
* Patients with rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption
* Lactating and pregnant women.
* Clinically significant abnormalities on physical examination, vital signs or laboratory tests at Visit 0 which in the opinion of the Investigator could interfere with the study procedures or endpoints evaluation.
* Suspicious or confirmed COVID-19 infection at time of screening visit.
* History of cervical, thoracic, or lumbosacral pain for ≥75% of the time in the last year, or of any other Low Back Pain episode in the last 3 months that required pharmacological treatment with an opioid analgesic.
* Patients with:

  * serious spinal pathology; spinal surgery in the year prior to screening or history of more than one spinal surgery; history of severe lumbar spinal stenosis; ankylosing spondylitis; lumbosciatalgia; herniated disc or radiculopathy; severe arthritis and osteoporosis; muscular diseases, such as myositis, poliomyelitis, muscular dystrophy and myotonia; fibromyalgia; myasthenia grave; fracture or recent history of violent trauma of the back; structural deformity of the back;
  * history of hypersensitivity to aspirin or any other non-steroidal anti-inflammatory drugs; suspicion of inflammatory, infective or neoplastic cause of pain; non- specific back symptoms related to abdominal, pelvic or thoracic pathology sensory and/or motor deficits in lower extremities;
  * history of gastroduodenal ulcer or bleeding;
  * history of severe cardiac, hepatic or renal insufficiency;
  * current anticoagulant therapy;
  * previous treatment with anticoagulants in the seven days before the screening visit;
  * concomitant use of physical or alternative therapies to treat current episode of pain;
  * local steroid injection for any reasons within previous 30 days;
  * alcohol or drug-addition or abuse;
  * cancer, not in remission or in remission less than 1 year;
  * active influenza or other viral syndrome; immunosuppression; systematically unwell; unexplained significant weight loss;
  * widespread neurological symptoms (including cauda equina syndrome) or any brain disease; ever suffered from any brain damage or have been in a coma; epilepsy or seizure;
  * active or suspected oesophageal, gastric, pyloric channel, or duodenal ulceration, or bleeding in the last 30 days;
  * blood-formation disturbance;
  * renal and/or hepatic failure;
  * acute hepatitis;
  * acetylsalicylic acid-triggered asthma;
  * history of asthma;
  * glucose-6-phosphate dehydrogenase-deficient patients; glutathione deficiency, dehydration, chronic malnutrition; anaemia.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the area under the pain intensity difference-versus-time curve of Low Back Pain scores up to 3 days of treatment | From Day 1 up to Day 3 (±1)
  The pain intensity difference will be considered to be the difference in VAS pain intensity between one time-point and the baseline. The sum of the pain intensity differences (SPID) will be the sum of the average of two consecutive pain intensity differences multiplied by the time-interval between two time points.

SECONDARY OUTCOMES:
Change in Visual Analogue Scale 0-10 cm (100 mm) | Day 0 and Day 8 (±1)
  Change in Visual Analogue Scale score at baseline (Visit 0) and at the end of study (Visit 2).The Visual Analogue Scale consists of a continuous horizontal line of 10 cm (100 mm) in length, on a piece of paper, with ends labelled as the extremes of pain, from 0 (left side): "no pain", to 10 (right side): "pain as bad as it could be". Patients will be asked to place a line with a pen perpendicular to the VAS line and intersecting the VAS line at the point that represents their current pain intensity.
Change from baseline up to the end of the study in Visual Analogue Scale 0-10 cm (100 mm) score. | From Day 0 to Day 8 (±1)
  Change from baseline up to the end of the study in VAS score, assessed at baseline (Visit 0) and Visit 2, and daily recorded in the patient diary during the whole home-stay period
Change from baseline up to the end of the study in the hand-to-floor distance | Day 0, Day 4 and Day 8 (±1)
  Change from baseline up to the end of the study in the hand-to-floor distance assessed at Visits 0, 1 and 2, measured by a cm graduated bar.
  The Hand-to-floor-distance, also called fingertip-to-floor test or mobility assessment, is a test to evaluate the mobility of both the whole spine and the pelvis in the overall motion of bending forward.
  The Investigator will ask the patient to stay erect on a platform 20-cm high with shoes removed and feet together. The patient will be asked to bend forward as far as possible and try to touch the floor with his/her fingers, while maintaining the knees, arms, and fingers fully extended. The vertical distance between the tip of the middle finger and the platform will be measured through a simple cm graduated bar (0 value at floor). The vertical distance between the platform and tip of the middle finger is positive when the subject does not reach the platform and negative when he/she can go further.
Change from baseline up to the end of the study in the in the degree of improvement in the functional disability | Day 0, Day 4 and Day 8 (±1)
  Change from baseline up to the end of the study in the in the degree of improvement in the functional disability, assessed at Visits 0, 1 and 2, measured by the Oswestry Disability Index (ODI).
  The Oswestry Disability Indexcontains 10 sections: (1) pain intensity, (2) personal care (washing/dressing), (3) lifting, (4) walking, (5) sitting, (6) standing, (7) sleeping, (8) sex life (if applicable), (9) social life, (10) travelling.
  Each section contains six statements that are scored from 0 (minimum degree of difficulty in that activity) to 5 (maximum degree of difficulty): if the first statement is marked, the section score is=0; if the last statement is marked, it is=5.
  The total score is the Oswestry Disability Index score and is obtained by summing up the scores of all sections, giving a maximum of 50 points.
  The final score is expressed as a percentage with the following formula: (total score/ (5 × number of questions answered) × 100%.
Change in the patients' global impression | Day 4 and Day 8 (±1)
  Change in the patients' global impression at Visits 1 and 2, measured by the Patients' Global Impression of Change (PGIC) scale.The patient will give the evaluation about his/her rating of overall improvement (if any) relative to a baseline state at the beginning of the treatment, according to the PGIC 7-point scale (Hurst and Bolton, 2004):
  1. No change (or condition has got worse)
  2. Almost the same, hardly any change at all
  3. A little better, but no noticeable change
  4. Somewhat better, but the change has not made any real difference
  5. Moderately better and a slight but noticeable change
  6. Better and a definite improvement that has made a real and worthwhile difference
  7. A great deal better and a considerable improvement that has made all the difference
Change in the clinical global impression | Day 4 and Day 8 (±1)
  Change in the clinical global impression at Visits 1 and 2, measured by the Clinical Global Impression-Improvement (CGI-I) scale.
  The Clinical Global Impression-Improvement (CGI-I) scale provides an overall clinician-determined summary evaluation of the treatment. the results in the appropriate source documents and on eCRF.
  The Investigator will assign a score based on how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the treatment, according to the following 7-point scale (Guy, 1976):
  1. Very much improved since the initiation of treatment
  2. Much improved
  3. Minimally improved
  4. No change from the initiation of treatment
  5. Minimally worse
  6. Much worse
  7. Very much worse since the initiation of treatment
Monitoring the frequency of adverse events | 8 (±1) days
  Safety will be assessed by monitoring the frequency of adverse events in each treatment group.
  AEs will be summarized using the total number of AEs, the total number and percentage of patients who experienced an AE, and the number and percentage of patients who experienced an AE within each System Organ Class (SOC) and by preferred term.

CONTACTS AND LOCATIONS:
Locations (11):
- Italy (3):
  - Università degli Studi della Campania "Luigi Vanvitelli", Caserta, CE
  - Azienda Ospedaliera Universitaria Policlinico G.Rodolico, Catania
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- Poland (8):
  - In-Vivo sp z o. o., Bydgoszcz
  - Przychodnia "Przy Szapitalu", Bydgoszcz
  - Zespół Porani Specjalistycznych Reumed Filia nr 1 Wallenroda, Lublin
  - Centrum Medyczne Pratia Poznan, Skorzewo
  - Nasz Lekarz Przychodnie Medyczne, Torun
  - Centrum Medyczne AstiMed, Warsaw
  - Centrum Medyczne PRATIA, Warsaw
  - Centrum Medyczne Reuma Park, Warsaw